CLINICAL TRIAL: NCT02514681
Title: A Randomized, Open-label Phase III Trial to Evaluate the Efficacy and Safety of Pertuzumab Retreatment in Previously Pertuzumab, Trastuzuamb and Chemotherapy Treated Her2-Positive Metastatic Advanced Breast Cancer
Brief Title: A Phase III Trial of Pertuzumab Retreatment in Previously Pertuzumab Treated Her2-Positive Advanced Breast Cancer
Acronym: PRECIOUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Breast Cancer Research Group (Other)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JBCRG-M05
Record Dates: First submitted 2015-07-28; First posted 2015-08-04 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: HER2-positive Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab; Docetaxel; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Vinorelbine; eribulin; Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Trastuzumab + chemotherapy (Active Comparator): Trastuzumab + chemotherapy Chemotherapy regimen is chosen from the following; Docetaxel, Paclitaxel, nab-paclitaxel ,Vinorelbine, Eribulin, Capecitabine or Gemcitabine
  Interventions: Drug: Trastuzumab; Drug: Docetaxel; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Vinorelbine; Drug: Eribulin; Drug: Capecitabine; Drug: Gemcitabine
- Trastuzumab+ pertuzumab + chemotherapy (Experimental): Trastuzumab+ pertuzumab + chemotherapy Chemotherapy regimen is chosen from the following; Docetaxel, Paclitaxel, nab-paclitaxel, Vinorelbine, Eribulin, Capecitabine or Gemcitabine
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Docetaxel; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Vinorelbine; Drug: Eribulin; Drug: Capecitabine; Drug: Gemcitabine

INTERVENTIONS:
Drug: Trastuzumab
  Other Names: Herceptin
Drug: Pertuzumab
  Other Names: Perjeta
  Arms: Trastuzumab+ pertuzumab + chemotherapy
Drug: Docetaxel
  Other Names: Taxotere
Drug: Paclitaxel
  Other Names: Taxol
Drug: Nab-paclitaxel
  Other Names: Abraxane
Drug: Vinorelbine
  Other Names: Navelbine
Drug: Eribulin
  Other Names: Halaven
Drug: Capecitabine
  Other Names: Xeloda
Drug: Gemcitabine
  Other Names: Gemzar

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pertuzumab, trastuzumab and chemotherapy as a pertuzumab retreatment compared to trastuzumab and chemotherapy in locally advanced or metastatic breast cancer patients for previously treated with pertuzumab

DETAILED DESCRIPTION:
The American Society of Clinical Oncology (ASCO) Clinical Practice Guidelines recommend the use of pertuzumab, trastuzumab and taxane as first-line treatment for patients with MBC. As a second-line treatment, trastuzumab emtansine (T-DM1) is also recommended. After a pertuzumab-containing regimen and T-DM1, other HER2-targeted therapeutic regimens, including lapatinib-containing regimens and trastuzumab plus chemotherapy, are recommended as third-line treatments and beyond. However, continual pertuzumab use for progression after a pertuzumab-containing regimen and retreatment with pertuzumab are unclear based on evidence.

The efficacy and the safety of two distinct modalities of a trastuzumab plus pertuzumab-containing regimen after pertuzumab use should be assessed in MBC: continual treatment and retreatment. However, it is clinically difficult to examine the efficacy of continual treatment with a trastuzumab plus pertuzumab-containing regimen because of several circumstances including the results of the MARIANNE study.

In addition, it is also important to evaluate the usefulness of retreatment with a pertuzumab-containing regimen. Continual pertuzumab treatment for progression after pertuzumab treatment is not same as pertuzumab retreatment. HER2-HER3-signaling suppressed by pertuzumab-containing regimens could potentially be restored by anti-HER2 therapy without pertuzumab. Pertuzumab retreatment could potentially re-suppress HER2-HER3-signaling. Therefore, Pertuzumab retreatment can be more effective than trastuzumab-containing treatment without pertuzumab.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed invasive breast cancer
2. A confirmed HER2-positive status assessed by means of immunohistochemical analysis (with 3+ indicating positive status) and/or in situ hybridization (with an amplification ratio > 2.0 indicating positive) by each institute
3. History of pertuzumab and trastuzumab-containing chemotherapy for locally advanced and metastatic breast cancer(2 or 3 regimen as previous chemotherapy regimen for locally advanced or metastatic breast cancer). The latest regimen before enrollment dose not include pertuzumab.
4. Patients have measurable and/or non-measurable disease according to RECIST ver1.1.
5. Female patients and aged ≥ 20 years.
6. Left Ventricular Ejection Fraction (LVEF) > 50% at baseline (within 28 days before enrollment) as determined by either ECHO or MUGA
7. Eastern Cooperative Oncology Group performance status of 0,1 or 2.
8. Life expectancy of patients is expected at least 3 months.
9. Signed and written informed consent (approved by the Institutional Review Board or Independent Ethics Committee) is obtained before any study procedure.

Exclusion Criteria:

1. History of chemotherapy > 4 regimen for locally advance or metastatic disease except for cancer chemotherapeutic agent-free treatment regimen (eg, hormonal therapy alone, combination with hormonal therapy and trastuzumab and anti-HER2 therapy alone).
2. Persistent Grade >3 non-hematologic toxicity according to NCI-CTCAE v4.0-JCOG resulting from previous therapy at the time of enrollment.
3. Symptomatic or uncontrolled central nervous system metastases.
4. Multiple malignancies without history of breast cancer(within 10 years if invasive breast cancer and within 5 years if malignancies except invasive breast cancer)
5. History of exposure to the following cumulative doses of anthracyclines:

   * doxorubicin or liposomal doxorubicin > 360 mg/m2
   * epirubicin > 720 mg/m2
   * mitoxantrone > 100 mg/m2
   * If more than 1 anthracycline has been used, then the cumulative dose must not exceed the equivalent of 360 mg/m2 of doxorubicin.
6. Current uncontrolled hypertension (systolic > 150 mmHg and/or diastolic > 100 mmHg) or unstable angina.
7. History of CHF of any New York Heart Association criteria, or serious cardiac arrhythmia requiring treatment (exception, atrial fibrillation, paroxysmal supraventricular tachycardia).
8. History of myocardial infarction within 6 months of enrollment.
9. Dyspnea at rest due to complications of advanced malignancy.
10. Inadequate organ function, as determined by the following laboratory results, within 28 days before enrollment:

    * Absolute neutrophil count < 1,500/mm3
    * Platelet count < 100,000/mm3
    * Hemoglobin < 8.0 g/dL
    * Total bilirubin > 2.0 mg/dL, unless the patient has documented Gilbert's syndrome
    * Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 100IU /L with the following exception (If considered that the liver dysfunction due to liver metastases > 200 IU/L, or 100 < , ≤200 IU/L with serum albumin < 2.5 g/dL)
    * Serum creatinine value > 2.0 mg/dL or 177 μmol/L
11. Current severe uncontrolled systemic disease(eg. Clinically significant cardiovascular, pulmonary and metabolic disease*, disorder of wound healing, ulcer and fracture)

    *If gemcitabine is planned to be selected as a combination chemotherapeutic agent,patients who has symptomatic interstitial pneumonia or pulmonary fibrosis on chest X-ray should be excluded.
12. Uncontrolled malignancy-associated hypercalcemia syndrome under bisphosphonates or denosumab treatment.
13. Radiation related grade >2 adverse event within 14 days before enrollment.
14. Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of need for major surgery during the course of study treatment.
15. Pregnant woman or positive pregnancy test.
16. Nursing woman
17. History of receiving any investigational treatment within 28 days before enrollment.
18. Current known and active infection with human immunodeficiency virus, hepatitis B virus or hepatitis C virus.
19. Receipt of intravenous antibiotics for infection within 14 days before enrollment.
20. Current chronic daily treatment (continuous for > 3 months) with corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids.
21. Known hypersensitivity to pertuzumab or trastuzumab without infusion reaction related to these drugs
22. Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (assessed by investigators) | 4 years

SECONDARY OUTCOMES:
Progression-free survival (assessed by independent review) | 4 years
PFS in patients treated with trastuzumab emtansine (T-DM1) as the latest regimen | 4 years
Response rate | 4 years
Duration of response, Overall survival | 4 years
Patient-reported-outcome | 4 years
  Difference in terms of patient-reported outcome (PRO) between standard group and Pertuzumab treated group FACT-G, FACT-B and EQ-5D are used as assessment tools for PRO.
Safety assessed by Incidence/Grade of Serious Adverse Events (SAEs), Pertuzumab-specific adverse events, laboratory abnormalities Percentage and number of subjects who discontinued for adverse event. | 4 years
  Safety for HER2-positive locally advanced or metastatic breast cancer subjects who were previously treated with Pertuzumab
Biomarkers | 4 years
  To find Prognostic and predictive biomarker markers for patients receiving anti-HER2 treatment. Changes in immunologic markers on peripheral blood mononuclear cells determined by flow cytometry after anti-HER2 treatment Changes in tumor-derived gene mutations (e.g. PIK3CA, APOBEC3, CDH1…etc.) in ctDNA after anti-HER2 therapy Changes in proteins (e.g. HER2, HER3…etc.) and micro RNAs expression in extracellular vesicle after anti-HER2 therapy Changes in glycans and proteins expression in the plasma after anti-HER2 therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroji Iwata, MD, PhD, Principal Investigator — Aichi Cancer Center Hospital; Yutaka Yamamoto, MD, PhD, Principal Investigator — Kumamoto University Hospital
Locations (3):
- Japan (3):
  - Aichi Cancer Center, Chikusa-ku, Aichi-ken
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Japan Breast Cancer Research Group, Chuo-ku, Nihonbashi, Koami-cho, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee-Hoeflich ST, Crocker L, Yao E, Pham T, Munroe X, Hoeflich KP, Sliwkowski MX, Stern HM. A central role for HER3 in HER2-amplified breast cancer: implications for targeted therapy. Cancer Res. 2008 Jul 15;68(14):5878-87. doi: 10.1158/0008-5472.CAN-08-0380. PMID 18632642
- [Background] Baselga J, Cortes J, Kim SB, Im SA, Hegg R, Im YH, Roman L, Pedrini JL, Pienkowski T, Knott A, Clark E, Benyunes MC, Ross G, Swain SM; CLEOPATRA Study Group. Pertuzumab plus trastuzumab plus docetaxel for metastatic breast cancer. N Engl J Med. 2012 Jan 12;366(2):109-19. doi: 10.1056/NEJMoa1113216. Epub 2011 Dec 7. PMID 22149875
- [Background] Giordano SH, Temin S, Kirshner JJ, Chandarlapaty S, Crews JR, Davidson NE, Esteva FJ, Gonzalez-Angulo AM, Krop I, Levinson J, Lin NU, Modi S, Patt DA, Perez EA, Perlmutter J, Ramakrishna N, Winer EP; American Society of Clinical Oncology. Systemic therapy for patients with advanced human epidermal growth factor receptor 2-positive breast cancer: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2014 Jul 1;32(19):2078-99. doi: 10.1200/JCO.2013.54.0948. Epub 2014 May 5. PMID 24799465
- [Background] Perez EA, Barrios C, Eiermann W, Toi M, Im YH, Conte P, Martin M, Pienkowski T, Pivot X, Burris H 3rd, Petersen JA, Stanzel S, Strasak A, Patre M, Ellis P. Trastuzumab Emtansine With or Without Pertuzumab Versus Trastuzumab Plus Taxane for Human Epidermal Growth Factor Receptor 2-Positive, Advanced Breast Cancer: Primary Results From the Phase III MARIANNE Study. J Clin Oncol. 2017 Jan 10;35(2):141-148. doi: 10.1200/JCO.2016.67.4887. Epub 2016 Nov 7. PMID 28056202
- [Derived] Yamamoto Y, Iwata H, Saji S, Takahashi M, Yoshinami T, Ueno T, Toyama T, Yamanaka T, Takano T, Kashiwaba M, Tsugawa K, Hasegawa Y, Tamura K, Tada H, Hara F, Fujisawa T, Niikura N, Taira N, Morita S, Toi M, Ohno S, Masuda N. Pertuzumab Retreatment for Human Epidermal Growth Factor Receptor 2-Positive Locally Advanced/Metastatic Breast Cancer (PRECIOUS Study): Final Overall Survival Analysis. J Clin Oncol. 2025 May 10;43(14):1631-1637. doi: 10.1200/JCO-24-01673. Epub 2025 Jan 24. PMID 39854662